CLINICAL TRIAL: NCT03722628
Title: The Assesment of Matrix Metalloproteinase-1 Genotypes Polymorphism as a Risk Factor for Hepatocellular Carcinoma in Chronic Hepatitis C Patients With Liver Cirrhosis
Brief Title: The Assesment of MMP-1 Genotypes Polymorphism as a Risk Factor for HCC in Chronic HCV Patients With LC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HMHassouna, Assistant Lecturer, Assiut University
Other Study IDs: MMP-1 in HCC
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- HCC with TTT: Blood sample from all HCC patients who recieved antiviral treatment for HCV will be taken to detect the MMP1-genotype polymorphism in those patients and the effect of treatment on this polymorphism.
  Interventions: Diagnostic Test: MMP1 genotypes polymorphism
- HCC without TTT: Blood sample from all HCC patients who didnot recieve antiviral treatment for HCV will be taken to detect the MMP1-genotype polymorphism in those patients and the effect of treatment on this polymorphism.
  Interventions: Diagnostic Test: MMP1 genotypes polymorphism
- LC with TTT: Blood sample from all LC patients who recieved antiviral treatment for HCV will be taken to detect the MMP1-genotype polymorphism in those patients and the effect of treatment on this polymorphism.
  Interventions: Diagnostic Test: MMP1 genotypes polymorphism
- LC without TTT: Blood sample from all LC patients who didnot recieve antiviral treatment for HCV will be taken to detect the MMP1-genotype polymorphism in those patients and the effect of treatment on this polymorphism.
  Interventions: Diagnostic Test: MMP1 genotypes polymorphism
- Healthy control: MMP1-genotype polymorphism will be applied on those healthy people to detect which type of mutation occur in healthy rather than diseased.
  Interventions: Diagnostic Test: MMP1 genotypes polymorphism

INTERVENTIONS:
Diagnostic Test: MMP1 genotypes polymorphism — Determination of MMP-1 gene polymorphism By PCR amplification followed by restriction Fragment length polymorphism (RFLP) and gel electrophoresis

SUMMARY:
Egypt is an endemic area of HCV.Cirrhosis and HCC are the most serious complications of chronic HCV infection.Some studies noted that the risk of HCC increased 17-fold among HCV-infected patients compared with anti-HCV negative controls.

Many studies demonstrate that direct antiviral therapy seems to accelerate the development of HCC, soon after the end of treatment, in those patients at higher risk of HCC occurrence or recurrence; and preliminary reports seem to indicate that HCC developed after direct antiviral therapy has more aggressive features. These findings clearly indicate the need for aggressive and close monitoring of cirrhotic patients during and after antiviral treatment, to detect and treat HCC at their earliest occurrence.

Genetic variation plays a key role in HCC susceptibility and development of the disease.Genotype distribution frequency data can be used to map single nucleotide polymorphism (SNP) diversity in a population and to examine the risk and development of specific diseases.Many reports indicate an association between SNPs in certain genes and the susceptibility and clinicopathological status of HCC.

MMP-1 is an endogenous peptide enzyme that is most widely expressed in interstitial collagenase,which can degrade the extracellular matrix surrounding tumor cells. It is involved in many stages of tumorigenesis, in angiogenesis, and in suppression of tumor cell apoptosis .

MMP-1 - 1607 1G/2G (rs1799750) contains a guanine insertion/deletion polymorphism at position - 1607 and is a functional (SNP) that can upregulate MMP expression. The association between the MMP-1 - 1607 1G/2G polymorphism and the emergence of several diseases including the risk for many cancers has been reported.

There are results suggest that MMP-1 is overexpressed in a large proportion of patients with HCC which correlated with the disease progression and poor clinical outcome. Furthermore, MMP-1 high expression proved to be a risk factor for tumor recurrence and independent molecular marker of prognosis in HCC and may become a novel target in the strategies for the prediction of tumor progression and prognosis of this disease.

Aim:

Is to asses:

The contribution of MMP-1-1607 genotype polymorphism to the risk of HCC on top of HCV.

The relationship between MMP-1-1607 gene polymorphism with HCC in patients who received antiviral treatment to HCV.

DETAILED DESCRIPTION:
This study is a case-control observational study to be done at Clinical pathology department, Assiut University hospital, Assiut University, Egypt. The control population comprised 20 healthy individuals with no liver infection. Patients will be subjected to a full history and thorough physical examination.The liver will be examined in all patients by local physical examination to detect possible abnormalities.The diagnosis of HCC cases include a combination of history, clinical examination ,radiological examination including ultrasound and triphasic computed tomography, Child-Pugh classification, and laboratory investigations including hepatitis C marker, irrespective of alpha-fetoprotein as it is positive in 30% of cases.

Neither patients nor controls had a history of other malignancy.The diagnosis of liver cirrhosis is based on clinical features, laboratory tests, abdominal ultrasound.

3-Exclusion criteria Exclude patients who had chronic hepatitis B virus infection by detecting HBsAg and core total, alcoholism, primary biliary cirrhosis, or autoimmune liver disease, decompensated liver cirrhosis on top of HCV .

4- Participants All individuals are subjected to the following:-

1. Full history taking including the history of taking antiviral drug,clinical examination, abdominal ultrasound.
2. Laboratory tests including:

   * Routine investigations: CBC,PT &PC,liver function tests.
   * Specific investigations: AFP level, serum level of MMP-1,Determination of MMP-1 gene polymorphism By PCR amplification followed by restriction Fragment length polymorphism (RFLP) and gel electrophoresis.

ELIGIBILITY:
Inclusion Criteria:

* The control popula¬tion comprised 20 healthy individuals with no liver infection. Patients will be subjected to a full history and thorough physical examination.
* The liver will be examined in all patients by local physical examination to detect possible abnormalities.
* The diagnosis of HCC cases include a combination of history, clinical examination ,radiological examination including ultrasound and triphasic computed tomography, Child-Pugh classification, and laboratory investigations including hepatitis C marker.

Exclusion Criteria:

* Exclude patients who had chronic hepatitis B virus infection by detecting HBsAg and core total IgG, alcoholism, primary biliary cirrhosis, or autoimmune liver disease, decompensated liver cirrhosis on top of HCV will be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hepatic patients ,males and females
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
The level of Matrix metalloprotinease-1 genotypes polymorphism in the study population | 48 hours
  detection by polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Ahmed Abdelhameed, MD, Study Chair — Assiut University; Mohammed Ismail Sedeek, MD, Study Chair — Assiut University; Neveen Abdelmonem Kamel, MD, Principal Investigator — Assiut University; Hadier Mostafa Hassouna, M.Sc, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shastry BS. SNP alleles in human disease and evolution. J Hum Genet. 2002;47(11):561-6. doi: 10.1007/s100380200086. PMID 12436191
- [Background] Wang B, Hsu CJ, Lee HL, Chou CH, Su CM, Yang SF, Tang CH. Impact of matrix metalloproteinase-11 gene polymorphisms upon the development and progression of hepatocellular carcinoma. Int J Med Sci. 2018 Apr 3;15(6):653-658. doi: 10.7150/ijms.23733. eCollection 2018. PMID 29725257